CLINICAL TRIAL: NCT00003405
Title: Treatment Protocol for Patients With Standard Risk Acute Myelogenous Leukemia and Its Variants: Induction Using High-Dose Cytarabine, Mitoxantrone and Ethyol; Consolidation With Cytarabine and Idarubicin and Maintenance With 13 Cis Retinoic Acid and Alpha Interferon
Brief Title: Combination Chemotherapy Plus Biological Therapy in Treating Patients With Acute Myelogenous Leukemia
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: No enrollment
Sponsor: Rush University Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000066413; P01CA075606 (NIH); RUSH-AML-9754; ALZA-RUSH-AML-9754; NCI-V98-1445
Record Dates: First submitted 1999-11-01; First posted 2004-05-24 (Estimated); Last update posted 2021-10-14 (Actual); Status verified 2021-10

CONDITIONS: Leukemia
Keywords: untreated adult acute myeloid leukemia; untreated childhood acute myeloid leukemia and other myeloid malignancies; adult acute erythroid leukemia (M6); adult acute myeloblastic leukemia without maturation (M1); adult acute myeloblastic leukemia with maturation (M2); adult acute myelomonocytic leukemia (M4); adult acute monoblastic leukemia (M5a); adult acute megakaryoblastic leukemia (M7); childhood acute myeloblastic leukemia without maturation (M1); childhood acute myeloblastic leukemia with maturation (M2); childhood acute myelomonocytic leukemia (M4); childhood acute monoblastic leukemia (M5a); childhood acute monocytic leukemia (M5b); childhood acute erythroleukemia (M6); childhood acute megakaryocytic leukemia (M7); adult acute monocytic leukemia (M5b)
MeSH Terms: conditions — Leukemia; Leukemia, Erythroblastic, Acute; Leukemia, Myeloid, Acute; Leukemia, Myelomonocytic, Acute; Leukemia, Monocytic, Acute; Leukemia, Megakaryoblastic, Acute | interventions — Interferon-alpha; Amifostine; Bromodeoxyuridine; Cytarabine; Idarubicin; Idoxuridine; Isotretinoin; Mitoxantrone

INTERVENTIONS:
Biological: recombinant interferon alfa
Drug: amifostine trihydrate
Drug: bromodeoxyuridine
Drug: cytarabine
Drug: idarubicin
Drug: idoxuridine
Drug: isotretinoin
Drug: mitoxantrone hydrochloride

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Biological therapies use different ways to stimulate the immune system and stop cancer cell from growing. Combining more than one chemotherapy drug with biological therapy may kill more cancer cells.

PURPOSE: Phase II trial to study the effectiveness of combination chemotherapy, isotretinoin, and interferon alfa in treating patients who have acute myelogenous leukemia.

DETAILED DESCRIPTION:
OBJECTIVES: I. Assess the efficacy of high dose cytarabine with mitoxantrone and amifostine as induction therapy for patients with previously untreated standard risk acute myelogenous leukemia (AML). II. Assess the effects of amifostine on the biology of AML cells in vivo in these patients. III. Determine whether there is a relationship between cytokine production before and during remission induction therapy and treatment outcome.

OUTLINE: Prior to treatment, patients undergo bone marrow aspirate and biopsy. On day -3, patients receive idoxuridine IV over 60 minutes followed immediately by a bone marrow aspirate and biopsy. Patients then receive amifostine IV over 5-7 minutes on the same day. Prior to chemotherapy on day 1, patient receive broxuridine IV over 60 minutes immediately followed by bone marrow aspirate and biopsy. Chemotherapy on day 1 consists of amifostine followed by cytarabine IV over 3 hours repeated every 12 hours and mitoxantrone IV over 1 hour immediately after the second infusion of cytarabine. This course is repeated on day 5 after another bone marrow biopsy and aspirate. Starting on day 6, patients receive amifostine 3 times a week until day 28 or beyond. Patients who respond to treatment continue on to receive three courses of consolidation therapy. Consolidation courses 1 and 3 consist of cytarabine continuous IV on days 1-7 and idarubicin IV over 30 minutes on days 1, 2, and 3. Consolidation course 2 consists of cytarabine IV over 75 minutes repeated every 12 hours for 4 days. Twenty-four hours after each course of consolidation therapy, patients receive isotretinoin orally every day and interferon alfa subcutaneously every other day. Isotretinoin and interferon alfa therapy are stopped 4 days prior to day 1 of the next course of consolidation therapy. Following recovery from course 3 of consolidation therapy, patients continue to receive isotretinoin/interferon alfa until relapse. Patients in complete remission after the 3 courses of consolidation therapy receive isotretinoin/interferon alfa for 3 years. Patients are followed every 3 months for the first year, then every 6 months for the next 2 years.

PROJECTED ACCRUAL: There will be 40-45 patients accrued into this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed previously untreated acute myelogenous leukemia (AML) FAB M1, M2, M4, M5, M6, or M7 No AML secondary to chemotherapy, radiation therapy, or toxic agents No history of myelodysplastic syndromes If possible, patient should be enrolled on protocol RUSH-CYL-9003

PATIENT CHARACTERISTICS: Age: 70 and under Performance status: 0-3 Life expectancy: Not specified Hematopoietic: Not specified Hepatic: Bilirubin greater than 2.0 mg/dL and no greater than 3.0 mg/dL allowed with 50% reduction in drug doses Renal: Creatinine less than 3.0 mg/dL Cardiovascular: No overt congestive heart failure No uncontrollable ventricular arrhythmias No uncontrollable hypertension If cardiac ejection fraction is less than 45% of predicted, an echocardiogram and a cardiac consult must be obtained to ascertain cardiac tolerance of anthracycline therapy Neurological: No cerebellar dysfunction Other: Fever, infection, or other complications of disease allowed Not pregnant or nursing Effective contraception required of all fertile patients

PRIOR CONCURRENT THERAPY: Biologic therapy: At least 2 weeks since prior interferon At least 2 weeks since prior hematopoietic growth factors (including erythropoietin) Chemotherapy: At least 2 weeks since prior chemotherapy Endocrine therapy: At least 2 weeks since prior steroids Radiotherapy: Not specified Surgery: Not specified Other: At least 2 weeks since prior retinoids

Ages: 0 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 1998-04; Primary Completion 1999-04; Study Completion 1999-04

CONTACTS AND LOCATIONS:
Overall Officials: Philip D. Bonomi, MD, Study Chair — Rush University Medical Center
Locations (4):
- United States (4):
  - Cook County Hospital, Chicago, Illinois
  - Rush Cancer Institute, Chicago, Illinois
  - Angelo P. Creticos, M.D. Cancer Center, Chicago, Illinois
  - Rush-Riverside Cancer Center, Kankakee, Illinois